CLINICAL TRIAL: NCT05069493
Title: Hiatal Hernia Repair by Tension-free Mesh Closure or Simple Suturing of the Diaphragmatic Hiatus. Long-term (>10 Years) Follow-up of a Randomized, Double-blind Clinical Trial
Brief Title: Long-term Follow-up After Hiatal Hernia Repair by Tension-free Mesh Closure or Simple Suturing
Status: Completed | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Collaborators: Ersta Hospital, Sweden (Other)
Responsible Party: Principal Investigator, Lars Lundell, professor, Karolinska University Hospital
Other Study IDs: PATCH2
Record Dates: First submitted 2021-09-26; First posted 2021-10-06 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: GERD; Hiatal Hernia; Dysphagia, Esophageal; Quality of Life
MeSH Terms: conditions — Gastroesophageal Reflux; Hernia, Hiatal; Deglutition Disorders | interventions — Melanocyte-Stimulating Hormones

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tension-free: Hiatal hernia repair by tension-free mesh closure
  Interventions: Procedure: mesh
- Suturing: Hiatal hernia repair by simple suturing of the diaphragmatic
  Interventions: Procedure: simple suturing

INTERVENTIONS:
Procedure: simple suturing — Hiatal hernia repair by simple suturing of the diaphragmatic
  Groups: Suturing
Procedure: mesh — Hiatal hernia repair by tension-free mesh closure
  Groups: Tension-free

SUMMARY:
10 years of follow-up after surgery for hiatal hernia by tension-free mesh closure or simple suturing.

DETAILED DESCRIPTION:
One-hundred and fifty-nine patients undergoing Nissen fundoplication for symptomatic gastro-oesophageal reflux disease (GORD), who had a concomitant hiatal hernia of > 2 cm axial length, were previously randomized to closure of the diaphragmatic hiatus with either crural sutures alone or tension-free closure with a non-absorbable mesh. Primary outcome variable was the incidence of radiologically verified recurrent hiatal hernia 3 years after the surgery and secondary outcomes were dysphagia score, reflux control and quality of life. The study showed no differences between the groups regarding hiatal hernia recurrence but higher dysphagia scores for solid food at 3 years in mesh group.

This study is a long-term follow-up (>10 years) after surgery for hiatal hernia by tension-free mesh closure or simple suturing.

ELIGIBILITY:
Inclusion Criteria:

-Patients available at the time of follow-up

Exclusion Criteria:

* Deceased
* Declined participation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who were included in the previous study (hiatal hernia repair by tension-free mesh closure or simple suturing) and are available for inclusion at the long-term follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Recurrent hiatal hernia | 10 years
  The incidence of radiologically verified recurrent hiatal hernia

SECONDARY OUTCOMES:
Dysphagia | 10 years
  Dysphagia for liquids and solids were recorded within a four-graded scale stating the frequency of dysphagia episodes with an arbitrary (empirical) cut off for clinical significance. The same dysphagia scoring was also used in a previous rct, from the same institution, comparing different types of antireflux procedures in open surgery.
Gastrointestinal symptom rating scale (GSRS) | 10 years
  A validated questionnaire containing five dimensions of abdominal symptoms (gastroesophageal reflux, abdominal pain, indigestion, obstipation and diarrhea
Quality of Life, physical and mental score: SF-36 | 10 years
  The Swedish version of the validated global Short Form -36 (SF-36) questionnaire was used and data are presented as physical and mental summary component scores (PCS and MCS, respectively)
Proton pump inhibitor (PPI) | 10 years
  Number of patients who report daily intake of PPI at the time of the follow up Use of PPI use of PPI

CONTACTS AND LOCATIONS:
Locations (1):
- Ersta Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Analatos A, Hakanson BS, Ansorge C, Lindblad M, Lundell L, Thorell A. Hiatal Hernia Repair With Tension-Free Mesh or Crural Sutures Alone in Antireflux Surgery: A 13-Year Follow-Up of a Randomized Clinical Trial. JAMA Surg. 2024 Jan 1;159(1):11-18. doi: 10.1001/jamasurg.2023.4976. PMID 37819652